CLINICAL TRIAL: NCT00980525
Title: Development of Inflammatory Disease Model Protein, Genetic and Microbial Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Janet Kinney, Associate Clinical Professor, University of Michigan
Other Study IDs: 2009-02
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plaque, saliva, and intraoral specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IL-1 genotype positive: There are three known IL-1 genes arranged in a cluster on human chromosome 2q13. Although the clinical application is still debatable, polymorphism in the IL-1 gene cluster was found to be associated with increased susceptibility to periodontal diseases. Conflicting studies demonstrate that a possible relationship between IL-1 genotype and clinical parameters of gingivitis may exist.This study will involve 15 subjects who are genotype positive and 15 subjects who are genotype negative.
- IL-1 genotype negative: There are three known IL-1 genes arranged in a cluster on human chromosome 2q13. Although the clinical application is still debatable, polymorphism in the IL-1 gene cluster was found to be associated with increased susceptibility to periodontal diseases. Conflicting studies demonstrate that a possible relationship between IL-1 genotype and clinical parameters of gingivitis may exist.This study will involve 15 subjects who are genotype positive and 15 subjects who are genotype negative.

SUMMARY:
The purpose of this study is to determine if certain levels of proteins lead to inflammation of the gums. One example of such proteins being studied is called Interleukin 1 (IL-1). This protein is found at higher levels in areas of inflammation. This type of study is called an experimental gingivitis study. It will involve stopping your routine oral health care for 21 days. If you qualify, you will receive a full dental cleaning at the beginning and end of the study. Approximately 30 patients will participate in this study at the Michigan Center for Oral Health Research (MCOHR).

DETAILED DESCRIPTION:
Gingivitis is a specific oral infectious disease that affects approximately 50% of the adult population on an average of 3 to 4 teeth. Although dental plaque is the primary etiology of most periodontal diseases, patients are not equally susceptible and do not respond similarly to professional care. Therefore, assessing the future risk of patients for developing gingivitis with possible subsequent progression to chronic periodontitis may help the clinician in elaborating a more accurate and suitable treatment plan for the patients and a better assessment of their prognoses. In fact, the prevention of plaque-induced gingivitis is still considered the first step in the maintenance of periodontal health.

Experimental gingivitis has been used widely to study the microbiology and the events that occur in the transition from a state of gingival health to inflammation. In a classical study by Löe and Theilade, periodontally healthy subjects were asked to cease all forms of oral hygiene for 3-4 weeks.

Studies of the levels of proinflammatory biomarkers have been of increased interest for the past decades. Since changes in the levels of these salivary biomarkers occur prior to clinical signs of gingivitis, their measurements may provide a more objective, earlier and accurate assessment of gingival inflammatory changes compared to the traditional bleeding and plaque indices.

Despite the clinical significance of gingivitis, little is know about the correlation between the levels of salivary biomarkers, the presence of periodontal pathogens and IL-1 polymorphism, and how this affect their susceptibility to gingivitis. If IL-1 polymorphism is indeed associated with increased levels of pro-inflammatory cytokines expression and the presence of specific periodontal pathogens, then screening for this polymorphism will be a valuable and necessary tool. As periodontal treatments, such as scaling and root planing, have been shown to be successful at decreasing the levels of IL-1 in the gingival crevicular fluid, a more aggressive treatment regimen may be warranted when the patient is genotype positive. If biomarkers in saliva and plaque biofilm can serve as accurate predictors of gingivitis, the ability for early detection of disease in patients is enhanced. Pro-inflammatory salivary biomarkers, specific pathogenic bacteria and genotype aid in establishing more accurate diagnostic and prognostic parameters of periodontal diseases, compared to current parameters (e.g. probing pocket depth, clinical attachment loss...) that reflect the history rather than the present and future status of disease. As a consequence, intervention can be initiated prior to irreversible tissue breakdown and oral health care costs may be reduced. Research efforts in the future should be directed toward the establishment of an affordable and practical chairside salivary test.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects between 18-40 years of age (throughout the study)
* Dentition with a minimum of 20 permanent teeth
* Mean score of less than or equal to 1 for plaque index, gingival index and papillary bleeding
* Compliance with all requirements in the study and signing the informed consent

Exclusion Criteria:

* Current smokers, smokers who quit less than one year ago, or a pack-year history of more than or equal to 10 (pack-years will be calculated by multiplying the number of years smoked by the average number of cigarette-packs smoked per day)
* Antibiotic therapy within 3 months of baseline or the need for antibiotics for infective endocarditis prophylaxis or other conditions
* Chronic medications known to affect the periodontal status (calcium antagonists, anticonvulsives, immunosuppressives, anti-inflammatory medications…)
* Pregnancy or lactating mothers
* Combined score of greater than 1 for plaque index, gingival index, and papillary bleeding at the screening visit
* Current orthodontic or periodontal treatments
* History of alcoholism or drug abuse
* Untreated carious lesions or defective restorations which could exacerbate during a period of oral hygiene abstinence
* Diseases of the immune system or any medical condition that may influence the outcome (diabetes, neurologic or psychiatric disorders, systemic infections…)
* New oral contraceptives users within 3 months of baseline or those planning on starting oral contraceptives during the study
* Depo-Provera contraceptive injection users

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will involve two groups: 15 subjects who are IL-1 genotype positive and 15 subjects who are IL-1 genotype negative. Potential participants will be recruited at the University of Michigan. A screening process will be performed by the study personnel to all potential participants to determine eligibility according to the inclusion and exclusion criteria. The prevalence of IL-1 genotype positive patients has been shown to be related to the patients' ethnic group. In Caucasians, the prevalence was found to be approximately 34% in non smokers. On the other hand, only about 2.3% of Asians and 26% of Hispanics were found to be IL-1 genotype positive. In order to limit ethnic variations, subjects in our study will be limited only to Caucasians.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to better understand the relationship between salivary proinflammatory biomarkers of gingivitis, the presence of specific bacteria and IL-1 polymorphism through experimental gingivitis. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kinney, RDH, MS, MS, Principal Investigator — University of Michigan, Department of Periodontics and Oral Medicine; William V Giannobile, DDS, DMed Sc, Study Director — University of Michigan Center for Oral Health Research
Locations (1):
- University of Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Loesche WJ. Clinical and microbiological aspects of chemotherapeutic agents used according to the specific plaque hypothesis. J Dent Res. 1979 Dec;58(12):2404-12. doi: 10.1177/00220345790580120905. PMID 41862
- [Background] Oliver RC, Brown LJ, Loe H. Periodontal diseases in the United States population. J Periodontol. 1998 Feb;69(2):269-78. doi: 10.1902/jop.1998.69.2.269. PMID 9526927
- [Background] Listgarten MA, Schifter CC, Laster L. 3-year longitudinal study of the periodontal status of an adult population with gingivitis. J Clin Periodontol. 1985 Mar;12(3):225-38. doi: 10.1111/j.1600-051x.1985.tb00920.x. PMID 3856578
- [Background] Kornman KS. Patients are not equally susceptible to periodontitis: does this change dental practice and the dental curriculum? J Dent Educ. 2001 Aug;65(8):777-84. PMID 11518250
- [Derived] Lee A, Ghaname CB, Braun TM, Sugai JV, Teles RP, Loesche WJ, Kornman KS, Giannobile WV, Kinney JS. Bacterial and salivary biomarkers predict the gingival inflammatory profile. J Periodontol. 2012 Jan;83(1):79-89. doi: 10.1902/jop.2011.110060. Epub 2011 May 12. PMID 21563952